CLINICAL TRIAL: NCT07362069
Title: E-cigarette Prevention and Emotion Regulation: Virtual Reality Intervention for Adolescents
Brief Title: A Virtual Reality Vaping Prevention Intervention for Adolescents
Status: Enrolling by invitation | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000039342; 1R01CA294027 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vaping
Keywords: vaping; prevention; emotion regulation; adolescents; virtual reality; intervention
MeSH Terms: conditions — Vaping; Emotional Regulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Focus Groups: Investigators will conduct focus groups with a sample of 8th-grade adolescents. To inform the conceptual model, investigators will ask students to describe perceptions about e-cigarettes and students' mental health needs in general, and how they perceive the link between the two constructs.
  Investigators will conduct interviews with 20 school staff, such as health teacher, school counselors, etc) to inform the implementation plan.

SUMMARY:
This study will examine E-Invite Only VR, a novel school-based universal e-cigarette prevention intervention that uses virtual reality (VR) to deliver prevention and emotion regulation skills-building content to middle school students in real-world classrooms. In Phase 1, investigators will conduct focus groups with adolescents and interviews with school staff to inform the development and implementation of the intervention.

DETAILED DESCRIPTION:
Investigators will conduct focus groups with adolescents. 4 focus groups will focus on collecting adolescents' perceptions about e-cigarettes and students' mental health needs in general, and how they perceive the link between the 2 constructs. Participants will also play E-Invite Only VR and then convene to share their thoughts and experiences. Participants will also fill out surveys including the System Usability Scale and the Gameplay Experience Questionnaire.

Staff will review and discuss the E-Invite Only VR implementation plan and respond to the Feasibility of Implementation Plan assessment during the interviews. Investigators will work with two populations: 1) Adolescents attending 8th grade in one of our partner schools, and 2) School staff employed by a partner school.

The target user for the E-Invite Only VR intervention is 8th grade students because the game is focused on prevention. Early adolescence is known to be a critical period for the risk of nicotine dependence and the transition between middle school and high school is a period when youth might be particularly likely to experiment with substances such as e-cigarettes.

Investigators will work with school staff to ensure the E-Invite Only VR intervention is feasible to implement in schools.

ELIGIBILITY:
School staff:

* employed by one of our partner schools
* could use the enhanced intervention with students OR work directly with students at risk for e-cigarette use/mental health concerns
* age greater than or equal to 18 years
* English speaking

  8th grade adolescents
* enrolled in 8th grade in one of our partner schools
* willing to engage in discussions about their experiences and perceptions related to e-cigarettes and mental health promotion
* English speaking

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The targeted study population is 8th grade adolescents and school staff (teachers, wellness coordinators, school counselors, and school psychologists) in participating schools.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the the Videogame | Immediately after the focus group and gameplay testing of the intervention, Day 1
  The Gameplay experience questionnaire, consisting of 11 items ranging from strongly disagree to strongly agree, will be used to assess adolescents' perception of the acceptability of the videogame intervention.
System Usability Scale | Immediately after the focus group and gameplay, Day 1
  The System Usability Scale (SUS), 10 items ranging from "strongly disagree" to "strongly agree" will be completed by adolescents and school staff to access the usability of the intervention.
Feasibility of Implementation | Immediately after interviews with school staff, Day 1
  Feasibility of Implementation, consisting of 5 items ranging from "Strongly disagree" to "strongly agree" will be used to assess feasibility of the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Investigators will make focus group data and associated documentation available to users only under a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will generally be available within one year of completion of the funded project period or upon acceptance of the first publication.
Access Criteria: Investigators will make focus group data and associated documentation available to users only under a data-sharing agreement that provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant, (2) a commitment to securing the data using appropriate computer technology, and (3) a commitment to destroying or returning the data after analyses are completed. Data will generally be available within one year of completion of the funded project period or upon acceptance of the first publication. Data will also be available through publications and presentations at scientific meetings. Findings will be published in scientific journals. All manuscripts that arise from this proposal will be submitted to PubMed Central.